CLINICAL TRIAL: NCT05613257
Title: A Randomized Controlled Trial Comparing Free-Hand Versus Distal Targeting Jig-Based for Distal Interlock Screw Placement
Brief Title: Distal Targeter vs Free-hand
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cedars-Sinai Medical Center (Other)
Collaborators: Stryker Nordic (Industry)
Responsible Party: Principal Investigator, Carol A. Lin, MD, Assistant Professor, Cedars-Sinai Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: STUDY00001778
Record Dates: First submitted 2022-10-31; First posted 2022-11-14 (Actual); Results first posted 2025-04-10 (Actual); Last update posted 2025-04-10 (Actual); Status verified 2025-04

CONDITIONS: Femur Fracture; Tibial Fractures; Nonunion of Fracture; Nonunion of Fracture of Tibia; Nonunion of Fracture of Femur (Diagnosis); Tibia Fracture
Keywords: femur fracture; tibia fracture; operative time; screw placement; jig
MeSH Terms: conditions — Femoral Fractures; Tibial Fractures; Fractures, Ununited; Disease

STUDY DESIGN:
Intervention Model Description: Patients will be randomly assigned to cohorts based on the operative technique used to treat their respective fractures.
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Free-hand/perfect circles (Active Comparator): Patients in this group will have interlocking screw placement using a free-hand, perfect circles technique.
  Interventions: Procedure: Free-hand/perfect circles technique
- Distal targeting jig (Experimental): Patients in this group will have interlocking screw placement using a proximally placed distal targeting jig
  Interventions: Device: Distal targeting jig

INTERVENTIONS:
Device: Distal targeting jig — Patients in this arm will have an assistive targeting device used for interlocking screw placement. The targeting device is attached to the nail proximally or distally (for antegrade or retrograde nailing, respectively) to guide screw placement through the other end of the intramedullary device.
  Arms: Distal targeting jig
Procedure: Free-hand/perfect circles technique — Patients in this arm will have no assistive targeting device use and the surgeon will use a free-hand technique for the placement of interlocking screws. With this technique, fluoroscopic images are taken such that the interlocking holes of the intramedullary device are "perfect circles" and indicate that a screw introduced in the same plane that the fluoroscopic image was taken would seat perpendicularly to the intramedullary device. This is the most commonly employed technique for interlocking screw placement through intramedullary devices.
  Arms: Free-hand/perfect circles

SUMMARY:
This study is a randomized controlled trial comparing the use of two different surgical techniques--free-hand versus distal targeting jig-based for distal interlock screw--placement and their effects on total operative time and intraoperative radiation exposure.

DETAILED DESCRIPTION:
Interlocking screw placement in intramedullary nailing of femoral and tibial shaft fractures improves rotational and length stability. However, free-hand perfect circle techniques can be technically challenging and may take up to an hour with increased radiation exposure to the surgeon and patient. Newer technologies aimed at reducing fluoroscope use such as electromagnetically-based aiming devices may increase the operative time. Proximally-based jigs have been shown to reduce fluoroscopy time in cadavers, however, have not been studied clinically. This study is a prospective, randomized controlled trial comparing a modern proximally-based distal targeting device and free-hand techniques for placement of interlocking screws in lower extremity nailing.

ELIGIBILITY:
Inclusion Criteria:

* 18 years old and above
* Undergoing intramedullary fixation of femur or tibia shaft for acute fracture or nonunion

Exclusion Criteria:

* Prior ipsilateral tibial or femoral nail
* Patients who cannot have interlocking screws placed
* Pregnant women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 89 (Actual)
Dates: Start 2022-10-31 (Actual); Primary Completion 2024-02-01 (Actual); Study Completion 2024-02-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Cedars Sinai Medical Center, Los Angeles, California, United States

REFERENCES:
- [Background] Maqungo S, Horn A, Bernstein B, Keel M, Roche S. Distal interlocking screw placement in the femur: free-hand versus electromagnetic assisted technique (sureshot). J Orthop Trauma. 2014 Dec;28(12):e281-3. doi: 10.1097/BOT.0000000000000125. PMID 24714403
- [Background] Miclau T, Holmes W, Martin RE, Krettek C, Schandelmaier P. Plate osteosynthesis of the distal femur: surgical techniques and results. J South Orthop Assoc. 1998 Fall;7(3):161-70. PMID 9781891
- [Background] Whatling GM, Nokes LD. Literature review of current techniques for the insertion of distal screws into intramedullary locking nails. Injury. 2006 Feb;37(2):109-19. doi: 10.1016/j.injury.2005.09.009. Epub 2005 Nov 28. PMID 16310192
- [Background] Program of Randomized Trials to Evaluate Pre-operative Antiseptic Skin Solutions in Orthopaedic Trauma (PREP-IT) Investigators; Slobogean GP, Sprague S, Wells J, Bhandari M, Rojas A, Garibaldi A, Wood A, Howe A, Harris AD, Petrisor BA, Mullins DC, Pogorzelski D, Marvel D, Heels-Ansdell D, Mossuto F, Grissom F, Del Fabbro G, Guyatt GH, Della Rocca GJ, Demyanovich HK, Gitajn IL, Palmer J, D'Alleyrand JC, Friedrich J, Rivera J, Hebden J, Rudnicki J, Fowler J, Jeray KJ, Thabane L, Marchand L, O'Hara LM, Joshi MG, Talbot M, Camara M, Szasz OP, O'Hara NN, McKay P, Devereaux PJ, O'Toole RV, Zura R, Morshed S, Dodds S, Li S, Tanner SL, Scott T, Nguyen U. Effectiveness of Iodophor vs Chlorhexidine Solutions for Surgical Site Infections and Unplanned Reoperations for Patients Who Underwent Fracture Repair: The PREP-IT Master Protocol. JAMA Netw Open. 2020 Apr 1;3(4):e202215. doi: 10.1001/jamanetworkopen.2020.2215. PMID 32259266
- [Derived] Stanley M, Huang K, Garlich J, Little M, Marecek G, Moon C, Vrahas M, Lin C. A Targeting Arm for Interlocking Screws Reduces Radiation Exposure: Results of a Prospective Randomized Controlled Trial. J Orthop Trauma. 2025 Dec 1;39(12):631-638. doi: 10.1097/BOT.0000000000003066. PMID 40892974

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Free-hand/Perfect Circles | Distal Targeting Jig
Started | 52 | 37
Completed | 33 | 29
Not Completed | 19 | 8

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Free-hand/Perfect Circles | Distal Targeting Jig | Total
Number analyzed (Participants) | 33 | 29 | 62
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 22 | 18 | 40
  >=65 years | 11 | 11 | 22
Age, Continuous [Median (Standard Deviation); unit: years] | 53 (23.32) | 43 (22.81) | 53 (22.90)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 17 | 35
  Male | 15 | 12 | 27
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 33 | 29 | 62

OUTCOME MEASURES:

1. Primary Outcome: Patient Radiation Exposure
Description: Number of fluoroscopic images taken intraoperatively for screw placement and cumulative radiation exposure (in grays)
Time Frame: During surgery: The first fluoroscopy shot for distal interlocking screw placement to final fluoroscopy shot confirming the final screw's placement
Measure: Mean (Standard Deviation); unit: images taken
Arm/Group | Free-hand/Perfect Circles | Distal Targeting Jig
Number analyzed (Participants) | 33 | 29
images taken | 47.03 (23.56) | 10.24 (10.63)

2. Primary Outcome: Total Screw Placement Time
Description: time taken to place interlocking screws
Time Frame: During surgery: the first fluoroscopy shot to localize the jig or obtain a perfect circle (start) to the last shot to confirm complete seating of the screw (end time)
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Free-hand/Perfect Circles | Distal Targeting Jig
Number analyzed (Participants) | 32 | 29
minutes | 14.87 (8.86) | 15.44 (14.33)

3. Primary Outcome: Measurement of Screw Placement Angle
Description: Correct screw placement is at a right (90-degree) angle from the intramedullary nail, through the interlocking screw hole
Time Frame: Intraoperatively (at end of surgery)
Population: Zero participants were analyzed as this data metric was not collected at the end of surgery in any of the participants as there was no reliable way to obtain this measurement.
Groups:
- Free-hand/Perfect Circles; Distal Targeting Jig: Zero participants were analyzed as this data metric was not collected.
Arm/Group | Free-hand/Perfect Circles | Distal Targeting Jig
Number analyzed (Participants) | 0 | 0

4. Primary Outcome: Amount of Cumulative Radiation Exposure (in Grays)
Description: Total radiation exposure during distal screw placement
Time Frame: as for outcome 1
Measure: Mean (Standard Deviation); unit: grays
Arm/Group | Free-hand/Perfect Circles | Distal Targeting Jig
Number analyzed (Participants) | 30 | 28
grays | 1.14 (1.19) | 1.51 (3.64)

ADVERSE EVENTS:
Time Frame: Adverse event data was collected for the first 30 days after surgery.
Arm/Group | Free-hand/Perfect Circles | Distal Targeting Jig
All-Cause Mortality (participants affected / at risk) | 0/33 | 0/29
Serious Adverse Events (participants affected / at risk) | 0/33 | 0/29
Other Adverse Events (participants affected / at risk) | 0/33 | 0/29

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-10-25): https://cdn.clinicaltrials.gov/large-docs/57/NCT05613257/Prot_SAP_002.pdf
  • Informed Consent Form (2023-10-25): https://cdn.clinicaltrials.gov/large-docs/57/NCT05613257/ICF_003.pdf